CLINICAL TRIAL: NCT01052298
Title: Randomized, Single-blinded, Placebo-controlled Study to Evaluate the Safety and Tolerability, the Pulmonary Deposition and Pharmacokinetics of Ciprofloxacin in Patients With Mild to Moderate Chronic Obstructive Pulmonary Disease (GOLD I - II), Following Inhalation of Ciprofloxacin PulmoSphere Inhalation Powder.
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of Inhaled Ciprofloxacin in Patients With Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13013; 2008-006770-14 (EudraCT Number)
Record Dates: First submitted 2009-10-15; First posted 2010-01-20 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Disease, Pulmonary
Keywords: Ciprofloxacin; Inhalation; Pharmacokinetics; Safety; Tolerability; COPD
MeSH Terms: conditions — Lung Diseases; Respiratory Aspiration; Pulmonary Disease, Chronic Obstructive | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro inhale, BAYQ3939)
- Arm 2 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro inhale, BAYQ3939)
- Arm 3 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro inhale, BAYQ3939)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro inhale, BAYQ3939) — 32.5 mg ciprofloxacin betaine corresponding to 50 mg Ciprofloxacin Pulmosphere inhalation powder will be given as an initial single dose application on day 00d.During the multiple dose phase (day 02d to 10d) the same dose will be given twice daily (bid) with a concluding single dose on 11d.
  Arms: Arm 1
Drug: Ciprofloxacin (Cipro inhale, BAYQ3939) — 32.5 mg ciprofloxacin betaine corresponding to 50 mg Ciprofloxacin Pulmosphere inhalation powder will be given as an initial single dose application on day 00d.During the multiple dose phase (day 02d to 10d) the same dose will be given three times daily (tid) with a concluding single dose on 11d.
  Arms: Arm 2
Drug: Ciprofloxacin (Cipro inhale, BAYQ3939) — 48.75 mg ciprofloxacin betaine corresponding to 75 mg Ciprofloxacin Pulmosphere inhalation powder will be given as an initial single dose application on day 00d.During the multiple dose phase (day 02d to 10d) the same dose will be given twice daily (bid) with a concluding single dose on 11d.
  Arms: Arm 3
Drug: Placebo — Placebo inhalation powder will be given as an initial single dose inhalation on 00d.During the multiple dose phase placebo will be given twice/three-times daily with a concluding single dose on day 11d.
  Arms: Arm 4

SUMMARY:
Objectives of the study are to investigate the safety, tolerability and levels of ciprofloxacin in the lung after single and multiple inhalative administration to patients with mild to moderate COPD (stage I-II according to GOLD Criteria).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COPD (Stage I or II according to the GOLD Classification), 35 years of age or older
* Airway obstruction with a post-bronchodilator Forced Expiratory Volume (FEV1) > or equal 50% of predicted normal and a post-bronchodilator FEV1 / Forced Vital Capacity (FVC) < 70%.
* Current or ex-smokers with a smoking history of more than 10 pack-years
* Body mass index (BMI) between 18 and 33 kg/m2
* Written informed consent to participate in the study after receiving adequate previous information and prior to any study specific procedures

Exclusion Criteria:

* Significant disease other than COPD as bronchial asthma, cystic fibrosis or clinically evident bronchiectasis
* Total blood eosinophil count >/=600/mm3.
* Thoracotomy with pulmonary resection
* Regular use of daytime oxygen therapy
* Completion of a pulmonary rehabilitation program in the six weeks prior to the pre-study examination or current participation in a rehabilitation program
* Hypersensitivity to the investigational drug or to other quinolones and/or to inactive constituents of the inhalation powder
* Hypersensitivity of the bronchial system to inhalation of nebulized drugs or saline solution
* Acute pulmonary exacerbation
* Patients with a history of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Concomitant inhalative therapy with antibiotics and/or concomitant systemic therapy with fluoroquinolones
* Oral beta-adrenergics, beta blockers
* Long acting anti-cholinergics within 2 weeks prior to pre-study examination
* Inhaled or oral steroids
* Methylxanthines: 24-hour washout of short-acting theophylline and 48-hour washout of long-acting theophylline prior to pre-study examination
* Antihistamines, antileukotrienes prescribed for asthma
* oral cromolyn sodium or oral nedocromil sodium

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Vital signs: evaluated by heart rate, blood pressure, clinical laboratory | Within 28 days after first treatment
Electrocardiogram: evaluated by shape and time intervals | Within 28 days after first treatment
Pulmonary function test evaluated by FEV1 | Within 28 days after first treatment
Pulse oximetry by peripheral oxygen concentration | Within 12 days after first treatment

SECONDARY OUTCOMES:
Determination of ciprofloxacin concentration in blood | Within 14 days after first treatment
Determination of ciprofloxacin concentration in urine | Within 14 days after first treatment
Determination of ciprofloxacin concentration in sputum | Within 14 days after first treatment
Determination of ciprofloxacin concentration in oral rinsing fluid | Within 7 days after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mannheim, Baden-Wurttemberg, Germany